CLINICAL TRIAL: NCT05395273
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of Cryocompression After Total Knee Arthroplasty (TKA)
Brief Title: Cryocompression After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-D0056
Record Dates: First submitted 2022-05-18; First posted 2022-05-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Cryotherapy Effect

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryocompression + standard therapy (Experimental): Participants received daily crycompression by the patient to their comfort level beside the standard therapy.
  Interventions: Device: Game Ready cryocompression
- Standard therapy (No Intervention): The standard therapy include the common physical therapy interventions, which are normally used in the hospital.

INTERVENTIONS:
Device: Game Ready cryocompression — Cryotherapy on the coldest tolerable level and intermittend compression on the knee
  Arms: Cryocompression + standard therapy

SUMMARY:
The overall aim of this study is to evaluate the effectiveness of a cryocompression device after total knee arthroplasty (TKA) compared to standard therapy.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of cryocompression after total knee arthroplasty (TKA) compared to a control group without cryocompression. The effect on the following parameters will be evaluated: knee and osteoarthritis outcome score (KOOS), patient satisfaction, knee girth, skin temperature, knee range of motion, morphine consumption, pain perception, the length of stay, the 10-metre walk test and the timed-up-and-go.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Diagnosed Arthritis of the Knee
* Planned implantation of a primary total knee arthroplasty by the Regionalspital Surselva AG

Exclusion Criteria:

* Decompensated hypertension in the affected area
* Acute inflammatory phlebitis in the affected area
* Patients with acute paroxysmal cold hemoglobinuria, or cryoglobulinemia
* Significant vascular disruption in the affected area
* History of pulmonary embolism or risk factors for deep vein thrombosis or pulmonary embolism in the affected area
* No increased venous or lymphatic return in the affected leg is desired due to e.g. carcinoma
* Raynaud's disease
* Hypersensitivity to cold
* Fear of cold/compression

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (preoperatively) Knee and Osteoarthritis Outcome Score (KOOS) at postoperatively (4th day) and 6 weeks after surgery | preoperatively, postoperatively (4th day) and 6 weeks after surgery
  A knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems
Change from Baseline (preoperatively) Range of motion at postoperatively (4th day) and 6 weeks after surgery | preoperatively, postoperatively (4th day) and 6 weeks after surgery
  Range of motion of the knee
Change from Baseline (preoperatively) Girth at postoperatively (4th day) and 6 weeks after surgery | preoperatively, postoperatively (4th day) and 6 weeks after surgery
  Knee girth
Change from Baseline (preoperatively) Timed up and Go at postoperatively (4th day) and 6 weeks after surgery | preoperatively, postoperatively (4th day) and 6 weeks after surgery
  A general physical performance test used to assess mobility, balance and locomotor performance
Change from Baseline (preoperatively) Skin temperature at postoperatively (4th day) and 6 weeks after surgery | preoperatively, postoperatively (4th day) and 6 weeks after surgery
  Skin temperature of the knee
Change from Baseline (preoperatively) Visual analogue scale at postoperatively (4th day) and 6 weeks after surgery | preoperatively, postoperatively (4th day) and 6 weeks after surgery
  To measure the intensity of pain
Change from Baseline (preoperatively) 10 Metre Walk Test at postoperatively (4th day) and 6 weeks after surgery | preoperatively, postoperatively (4th day) and 6 weeks after surgery
  To assess walking speed in meters per second over 10 metres
Change from Baseline (first day postperatively) Patient satisfaction at each day of hospitalisation | each day of hospitalisation
  To measure the patient satisfaction of the cryocompression therapy from 0 to 10
Consumption of morphine | 6 weeks after surgery
  Consumption of morphine in number of pills
Length of stay | 6 weeks after surgery
  Length of stay in the hospital in days

CONTACTS AND LOCATIONS:
Overall Officials: Ron Clijsen, PhD, Principal Investigator — University of Applied Sciences and Arts of Southern Switzerland
Locations (1):
- Fachhochschule Südschweiz, Landquart, Kanton Graubünden, Switzerland

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT05395273/Prot_SAP_000.pdf